CLINICAL TRIAL: NCT03415529
Title: Incidence of Hypercapnia and Impact of Arterial CO2 Tension on Management and Outcome in Patients With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Impact of Arterial CO2 Tension on Management and Outcome in Patients With Acute Hypoxemic Respirator Failure and ARDS
Acronym: CO2 LUNG SAFE
Status: Completed | Type: Observational
Sponsor: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: CO2LUNGSAFE
Record Dates: First submitted 2018-01-17; First posted 2018-01-30 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Acute Severe Respiratory Failure; Acute Respiratory Distress Syndrome
Keywords: Lung; ARDS; Acute Respiratory Syndrome; Prognosis; Outcome Research; Respiratory infection; Sepsis; Organ failure; Hypercapnia
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Tract Infections; Sepsis; Hypercapnia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 4500 patients with ARDS: This is a secondary analysis of data from the LUNG SAFE database to determine the impact of alterations in arterial carbon dioxide tensions in patients with ARDS.

SUMMARY:
There appears to be considerable variability in the approach physicians use to manage arterial carbon dioxide tensions, in patients in the early phases [first 48 hours] of ARDS (Acute hypoxemic respiratory failure and). A number of specific concerns exist, particularly the use of greater than needed inspired oxygen concentrations (potentially in 40% patients), and the proportion of hypocapnic patients in our cohort.

DETAILED DESCRIPTION:
This study will address a number of specific concerns, including:

1. the incidence of hypocapnia and hypercapnia;
2. the factors (e.g. ventilatory mode) contributing to hypocapnia and hypercapnia;
3. the impact of hypocapnia and hypercapnia on progression of ARDS, duration of ventilation, ICU stay, hospital stay and patient outcome;
4. the impact of pH (respiratory versus metabolic cause) on outcome variables.

LUNG SAFE was a prospective observational study. There was not patient intervention. The current analysis is a secondary analysis of this existing database.

Data will be abstracted form the database on all patients meeting the inclusion criteria for ARDS (during the first 2 days from AHRF onset) for the following variables: Patient's demographic characteristics (age, sex) and chronic comorbidities, Arterial PCO2, pH in first 48 hours, Data on P/F ratio over course of illness, Duration of ventilation, ICU stay, hospital survival in patients identified as being exposed to hypocapnia (pCO2 < or = to 30mmHg) and hypercapnia (PCO2 > or = to 45mmHg); Main ventilatory variables: mode of ventilation, tidal volume, respiratory.

Descriptive statistics will include proportions for categorical and mean (standard deviation) or median (interquartile range) for continuous variables, according the data distribution. The amount of missing data in the LUNG SAFE database is low so no assumptions will be made for missing data.

In order to investigate the relationship between PaCO2 and management factors, the investigators will stratify study population according the presence or absence of hypercapnia and will evaluate differences in management factors, using appropriate statistical tests. In detail, proportions will be compared using chi-squared or Fisher exact tests and mean values were compared using T-test or Wilcoxon rank sum test, as appropriate. Shapiro-Wilks test will be used to assess normality in data distribution. Moreover, they will perform univariate and multivariable logistic regression models using hypercapnia as dependent variable. Stepwise regression approach with significance alpha levels of 0.05 (both for entry and retention) will be used to establish a set of independent predictors. Odds ratios (ORs) and 95% confidence intervals (CIs) will be reported as measure of association.

They will assess the association of hypercapnia with different outcomes (ARDS progression, duration of mechanical ventilation, ICU and hospital stay and mortality) using generalized linear regression models (Poisson or Logistic regression models, according outcome distribution) and adjusting the relationship with all possible confounders identified with stepwise approach. Results will be reported as ORs, incidence rate ratios and corresponding 95% CI.

Particular attention will be given to the relationship and interaction between pH and PaCO2.

Survival analysis (Kaplan-Meier approach) will be used to estimate the time of liberation from invasive mechanical ventilation, of ICU and hospital discharge, and of hospital mortality within 28 days of AHRF onset in patients with and without hypercapnia. Differences in survival time will be assess by Log-Rank test.

ELIGIBILITY:
Inclusion Criteria:

* All patients meeting criteria for ARDS. Fulfillment of criteria for Acute Hypoxaemic respiratory failure (AHRF) and fulfillment of Berlin criteria for ARDS during the first two days after AHRF onset.

Exclusion Criteria:

* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who fulfilled clinical criteria for ARDS and Acute Hypoxaemic respiratory failure were recruited into the LUNG SAFE trial (NCT02010073) that was published in JAMA, 2016 Jul 19;316(3):347).
Sampling Method: Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence | LUNG SAFE was a prospective observational study. Patients were followed until hospital discharge or day 90, whichever came first
  The incidence of hypercapnia [i.e. PaCO2 > 45 mmHg] when ARDS arises

SECONDARY OUTCOMES:
Severity | LUNG SAFE was a prospective observational study. Patients were followed until hospital discharge or day 90, whichever came first
  The severity of hypercapnia [i.e. PaCO2 > 45 mmHg] when ARDS arises ARDS
Hypercapnia | LUNG SAFE was a prospective observational study. Patients were followed until hospital discharge or day 90, whichever came first
  Factors (e.g. ventilatory mode) contributing to hypercapnia in patients with ARDS
Hypercapnia | LUNG SAFE was a prospective observational study. Patients were followed until hospital discharge or day 90, whichever came first
  The impact of hypercapnia on outcome on the progression of ARDS
pH ((potential of hydrogen) | LUNG SAFE was a prospective observational study. Patients were followed until hospital discharge or day 90, whichever came first
  The impact of pH (respiratory versus metabolic cause) on outcome variables

CONTACTS AND LOCATIONS:
Overall Officials: John LAFFEY, Principal Investigator — National University of Ireland, Galway; Giacomo BELLANI, Principal Investigator — University of Milano-Bicocca (Monza, Italy)
Locations (1):
- Guy Marie FRANCOIS, Brussels, Belgium

REFERENCES:
- [Background] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Background] Laffey JG, Bellani G, Pham T, Fan E, Madotto F, Bajwa EK, Brochard L, Clarkson K, Esteban A, Gattinoni L, van Haren F, Heunks LM, Kurahashi K, Laake JH, Larsson A, McAuley DF, McNamee L, Nin N, Qiu H, Ranieri M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Correction to: Potentially modifiable factors contributing to outcome from acute respiratory distress syndrome: the LUNG SAFE study. Intensive Care Med. 2018 Jan;44(1):157-165. doi: 10.1007/s00134-017-4981-z. PMID 29138899
- [Background] de Prost N, Pham T, Carteaux G, Mekontso Dessap A, Brun-Buisson C, Fan E, Bellani G, Laffey J, Mercat A, Brochard L, Maitre B; LUNG SAFE investigators; ESICM trials group; REVA network. Etiologies, diagnostic work-up and outcomes of acute respiratory distress syndrome with no common risk factor: a prospective multicenter study. Ann Intensive Care. 2017 Dec;7(1):69. doi: 10.1186/s13613-017-0281-6. Epub 2017 Jun 19. PMID 28631088
- [Background] Laffey JG, Madotto F, Bellani G, Pham T, Fan E, Brochard L, Amin P, Arabi Y, Bajwa EK, Bruhn A, Cerny V, Clarkson K, Heunks L, Kurahashi K, Laake JH, Lorente JA, McNamee L, Nin N, Palo JE, Piquilloud L, Qiu H, Jimenez JIS, Esteban A, McAuley DF, van Haren F, Ranieri M, Rubenfeld G, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Geo-economic variations in epidemiology, patterns of care, and outcomes in patients with acute respiratory distress syndrome: insights from the LUNG SAFE prospective cohort study. Lancet Respir Med. 2017 Aug;5(8):627-638. doi: 10.1016/S2213-2600(17)30213-8. Epub 2017 Jun 15. PMID 28624388
- [Background] Dreyfuss D, Gaudry S, Madotto F, Laffey JG. Some remaining important questions after LUNG SAFE : Discussion of "Potentially modifiable factors contributing to outcome from acute respiratory distress syndrome: the LUNG SAFE study". Intensive Care Med. 2017 Apr;43(4):598-599. doi: 10.1007/s00134-017-4706-3. Epub 2017 Feb 17. No abstract available. PMID 28213623
- [Background] Laffey JG, Bellani G, Pham T, Fan E, Madotto F, Bajwa EK, Brochard L, Clarkson K, Esteban A, Gattinoni L, van Haren F, Heunks LM, Kurahashi K, Laake JH, Larsson A, McAuley DF, McNamee L, Nin N, Qiu H, Ranieri M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators and the ESICM Trials Group. Potentially modifiable factors contributing to outcome from acute respiratory distress syndrome: the LUNG SAFE study. Intensive Care Med. 2016 Dec;42(12):1865-1876. doi: 10.1007/s00134-016-4571-5. Epub 2016 Oct 18. PMID 27757516
- [Background] Bellani G, Laffey JG, Pham T, Madotto F, Fan E, Brochard L, Esteban A, Gattinoni L, Bumbasirevic V, Piquilloud L, van Haren F, Larsson A, McAuley DF, Bauer PR, Arabi YM, Ranieri M, Antonelli M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Noninvasive Ventilation of Patients with Acute Respiratory Distress Syndrome. Insights from the LUNG SAFE Study. Am J Respir Crit Care Med. 2017 Jan 1;195(1):67-77. doi: 10.1164/rccm.201606-1306OC. PMID 27753501
- [Background] Bellani G, Laffey JG, Pham T, Fan E; LUNG SAFE Investigators and the ESICM Trials Group. The LUNG SAFE study: a presentation of the prevalence of ARDS according to the Berlin Definition! Crit Care. 2016 Sep 9;20(1):268. doi: 10.1186/s13054-016-1443-x. No abstract available. PMID 27608629
- [Background] Bellani G, Pham T, Laffey J; LUNG-SAFE Investigators; ESICM Trials Group. Incidence of Acute Respiratory Distress Syndrome--Reply. JAMA. 2016 Jul 19;316(3):347. doi: 10.1001/jama.2016.6471. No abstract available. PMID 27434453